CLINICAL TRIAL: NCT04544020
Title: Changes in gUt micRobiota After Enteral Feeding (in Alcoholic Hepatitis)
Acronym: CREED
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019GA002
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Alcoholic Hepatitis
Keywords: gut microbiome; NG feeding
MeSH Terms: conditions — Hepatitis, Alcoholic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — stools
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- subjects: subjects with alcoholic hepatitis receiving NG feeding
  Interventions: Dietary Supplement: NG feeding

INTERVENTIONS:
Dietary Supplement: NG feeding — NG feeding

SUMMARY:
Drinking large amount of alcohol can cause damage to the liver. If the liver is severely injured by alcohol it can become very inflamed and this condition is called alcoholic hepatitis. Alcoholic hepatitis can be life threatening. There is no cure for alcoholic hepatitis. It is known that stop drinking and have good nutrition can help the liver to recover.

Infections are very common for people who suffer from alcoholic hepatitis. Sometimes these infection can be very severe. It is not always possible to find out where the infection is coming from. But the bacteria living in the bowel may move to other organs causing these infections and an illness like alcoholic hepatitis can cause "bad bacteria" to take over from "good bacteria" in the gut.

This study wants to understand the changes in the bacteria in the bowel of people who have an acute inflammation of the liver cause by alcohol (alcoholic hepatitis).

The investigators will take stool samples from patients admitted in the hospital with alcoholic hepatitis. The investigators will run tests on the stools that can find out which bacteria live in the bowel. Its is expected to find these bacteria to be different from the ones living in the bowel of healthy people. The investigators are interested to see if these bacteria change once the patients are given good nutrition using a small tube from the nose to the stomach. This type of nutrition is used routinely to help improve the liver in severe alcoholic hepatitis. The investigators will take some more stool sample from these patients after the nutrition through the tube has started to check how the bacteria change with nutrition.

Better tools to check the bacteria in the bowel are now available so this can help the investigators to understand better if changing bacteria in the bowel can help recovery in alcoholic hepatitis.

DETAILED DESCRIPTION:
Subjects admitted to hospital with a diagnosis of alcoholic hepatitis and who are planned to receive nasogastric feeding for at least 7 days will be eligible for the study.

A stool sample will be collected prior to commence enteral nutrition via nasogastric tube and analysed. Subsequently further stool samples will be collected and analysed at day 3 and day 7 after commencing nasogastric feeding.

DNA will be extracted from each of the samples, and bacterial 16S rRNA genes will be PCR amplified and sent for sequencing at the CGEBM using an Illumina MiSeq machine. This will generate at least 2 million paired end reads (2 x 300 bp), which will be assembled and analysed using the Mothur software platform.The investigators will also analyse the short chain fatty acids profiles within the stool samples using gas chromatography. Shannon Diversity Index will be used to assess the bacterial diversity and Pielou's index will be used to assess species evenness at each time point. Comparison between time points will be performed. Microbiota composition at the different time points will be assessed using Mothur software to detect if there are systematic changes to specific members of the gut microbiota during enteral feeding. Prevalence by different molecular methodologies will be assessed and the results from study patients will be compared with their baseline samples by Fisher's exact test.

Missing data will be handled using a missing indicator.

Subjects will be approached by the team in charge of the clinical care and option to enter the study will be offered. Information leaflet will be provided to the subject 24h before consenting and possibility to discuss with trial team.

Data will be collected by authorised members of trial team in a fit for purpose ad hoc password protected excel data base as eCRF. Source data will be electronic patient file or paper case notes. Source data of microbiome analysis will be computer report. Accuracy of data entry will be checked by a separate delegated member of the team. External monitoring occurs at a regular basis for clinical trial arrange by sponsor.

Patient confidentiality will be maintained at all time. No identifiable data will be collected. eCRF will be password protected and stored in encrypted hospital computer protected by password. consent or other paper documentation will be kept separate in locked cabinets within the premises of the hospital.

Adverse Events reporting will be performed by a competent and delegated member of staff, according to our sponsor standard operating procedure and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients: age 16 and above
* Diagnosis of alcoholic hepatitis confirmed by treating hepatologists and defined as:
* Bilirubin >80 umol/l
* Documented history of continuing alcohol harmful use
* ALT< 500 umol/L
* Clinical decision to start NG feeding and prospect to continue NG feeding >3 days

Exclusion Criteria:

* Age <16
* Hepatocellular carcinoma
* Pregnancy and breastfeeding
* Inability to provide informed consent
* Any reasons in the opinion of the investigator which can compromise participation in the trial or affect patient health

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - adults admitted to hospital. Diagnosis of alcoholic hepatitis. Expected to receive nasogastric feeding for at least 3 days.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
alteration of bacterial microbiome diversity and evenness following enteral feeding in alcoholic hepatitis | 7 days
  To understand how the gut microbiome changes in patients with AH following enteral feeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
we will plan to share all patient IPD, protocol including analysis plan

REFERENCES:
- [Background] Moreno C, Deltenre P, Senterre C, Louvet A, Gustot T, Bastens B, Hittelet A, Piquet MA, Laleman W, Orlent H, Lasser L, Serste T, Starkel P, De Koninck X, Negrin Dastis S, Delwaide J, Colle I, de Galocsy C, Francque S, Langlet P, Putzeys V, Reynaert H, Degre D, Trepo E. Intensive Enteral Nutrition Is Ineffective for Patients With Severe Alcoholic Hepatitis Treated With Corticosteroids. Gastroenterology. 2016 Apr;150(4):903-10.e8. doi: 10.1053/j.gastro.2015.12.038. Epub 2016 Jan 5. PMID 26764182
- [Background] Dubinkina VB, Tyakht AV, Odintsova VY, Yarygin KS, Kovarsky BA, Pavlenko AV, Ischenko DS, Popenko AS, Alexeev DG, Taraskina AY, Nasyrova RF, Krupitsky EM, Shalikiani NV, Bakulin IG, Shcherbakov PL, Skorodumova LO, Larin AK, Kostryukova ES, Abdulkhakov RA, Abdulkhakov SR, Malanin SY, Ismagilova RK, Grigoryeva TV, Ilina EN, Govorun VM. Links of gut microbiota composition with alcohol dependence syndrome and alcoholic liver disease. Microbiome. 2017 Oct 17;5(1):141. doi: 10.1186/s40168-017-0359-2. PMID 29041989
- [Background] Puri P, Thursz M. Intensive Enteral Nutrition in Alcoholic Hepatitis: More Food for Thought. Gastroenterology. 2016 Apr;150(4):803-5. doi: 10.1053/j.gastro.2016.02.061. Epub 2016 Feb 26. No abstract available. PMID 26924095